CLINICAL TRIAL: NCT02785484
Title: Randomized Controlled Trial Evaluating the Impact of Cigarette Pack Constituent Disclosures
Brief Title: Impact of Cigarette Pack Constituent Disclosures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-2430; P50CA180907 (NIH)
Record Dates: First submitted 2016-04-04; First posted 2016-05-27 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Cigarette Smoking Behavior
Keywords: Cigarette smoking; Smoking; Tobacco use
MeSH Terms: conditions — Cigarette Smoking; Smoking; Tobacco Use | interventions — Drug Labeling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Label with constituent disclosure message (Experimental)
  Interventions: Other: Label with constituent disclosure message
- Label with litter message (Other)
  Interventions: Other: Label with litter message

INTERVENTIONS:
Other: Label with constituent disclosure message — Labels with constituent disclosure messages that include text about chemicals in cigarette smoke and health effects of the chemicals will be applied to participants' cigarette packs on the right side (the Surgeon General's warning is on the left side). At the week 2 visit, participants' packs will be labeled with 1 of 3 disclosures selected at random; at the week 3 visit, they will get one of the 2 remaining disclosures selected at random, and at the week 4 visit they will get the remaining disclosure. Study investigators developed the text and design of these labels.
  Arms: Label with constituent disclosure message
Other: Label with litter message — Labels with litter messages that include text about littering cigarette butts will be applied to participants' cigarette packs on the right side (the Surgeon General's warning is on the left side). At the week 2 visit, participants' packs will be labeled with 1 of 3 litter messages selected at random; at the week 3 visit, they will get one of the 2 remaining litter message selected at random, and at the week 4 visit they will get the remaining litter message. Study investigators developed the text and design of these labels.
  Arms: Label with litter message

SUMMARY:
The purpose of this randomized controlled trial is to determine whether constituent disclosures on cigarette packs increase intentions to quit smoking. Previous studies have been informative, but they have evaluated candidate graphic warnings, not constituent disclosures. Furthermore, they typically expose participants to messages in controlled but artificial experimental settings for a short period of time, using much lower frequency and shorter duration of message exposure than found in the real world. This study addresses these issues by evaluating the impact of constituent disclosures by randomly assigning smokers to have their cigarette packs labeled with constituent disclosure messages or cigarette butt littering messages.

DETAILED DESCRIPTION:
Federal law requires the U.S. Food and Drug Administration (FDA) to disseminate information about tobacco constituents. The 2009 Family Smoking Prevention and Tobacco Control Act grants FDA broad authority to regulate tobacco products, including helping the public to better understand harmful and potentially harmful constituents (HPHCs) present in tobacco products and tobacco smoke. According to Section 206 of the Act, using the appropriate federal rulemaking channels and procedures, FDA may require disclosure of tobacco constituents if the disclosed information benefits public health and increases consumer awareness of the health consequences of tobacco products. This study will assess the impact of constituent disclosures on smokers' cigarette packs in a randomized control trial.

Recruitment: Smokers will first undergo screening online or call the study center to complete the screening questionnaire over the phone. Study staff will schedule eligible smokers for 5 in-person visits. For each of their 5 visits, smokers will be asked to bring the number of cigarettes they expect to smoke in an 8 day period.

Informed Consent: Prior to consenting smokers, research staff will visually inspect photo identification of smokers who report or appear to be under age 27. At the beginning of the first appointment, study personnel will explain the consent form and ask the smoker to read the form. Once the participant has finished reading the form, the study personnel member will ask the participant if he or she has any questions. Then both parties will sign the consent form and the participant will receive a copy of the consent form.

Randomization: At the week 2 visit, study personnel will randomly assign participants to one of the two study arms. The investigators will determine the randomization order a priori. Smokers have an equal chance of being randomized to have labels with constituent disclosure messages or labels with litter messages applied to their cigarette packs.

Assessment: Participants will complete 5 computer-based surveys during the study. The first appointment will take around 60 minutes and each subsequent visit will take around 30-45 minutes to complete. At all 5 visits, participants will complete a survey. At visits 2-4, participants' will have their cigarette packs labeled based on their condition. Cigarette packs will be tracked at all 5 study visits.

Detailed description of the intervention: Each week participants will bring in 8 days' of cigarettes (one extra day to provide a buffer in case of rescheduled appointments or smoking more than anticipated) for labeling and tracking. Additionally, they will bring in any unused labeled packs from the previous visit when applicable. While participants are taking the survey, research staff will count participants' cigarette packs. Study staff will mark packs with a code indicating the date of the visit and label them.

Participants randomized to the intervention arm will have labels with constituent disclosure messages applied to their cigarette packs during visits for weeks 2-4. Constituent disclosures that include text about chemicals in cigarette smoke and health effects of the chemicals will be applied to participants' cigarette packs as labels on the right side (the Surgeon General's warning is on the left side). At the week 2 visit, participants' packs will be labeled with 1 of 3 disclosures selected at random; at the week 3 visit, they will get one of the 2 remaining disclosures selected at random, and at the week 4 visit they will get the remaining disclosure. Study investigators developed the text and design of these labels. Participants assigned to the control arm will have labels with litter messages applied to the right side of their cigarette packs.

The investigators will instruct participants in both arms to smoke or not smoke as they normally would. The investigators will assess how many cigarettes participants smoked from packs previously brought to a visit and other sources to calculate intervention dose (% of cigarettes smoked from labeled packs). At the end of the study, participants will receive a list of cessation resources.

ELIGIBILITY:
Inclusion Criteria:

* Be 21 years or older
* Have smoked at least 100 cigarettes in his or her lifetime
* Currently smoke cigarettes every day or some days
* Currently smoke at least 7 cigarettes per week, on average
* Be able to read and speak English
* Be able to use a computer to take surveys
* Be able to attend 5 weekly appointments
* Be able to bring in 8 days' worth of cigarettes to each of the first 4 weekly appointments

Exclusion Criteria:

* Smokers who smoke exclusively roll-your-own cigarettes
* Pregnant women
* Smokers concurrently enrolled in any research studies about smoking or using other tobacco products
* Smokers who live in the same household as someone who has enrolled in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 784 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Quit intentions | 4 weeks
  The primary outcome is quit intentions measured at 4 weeks by survey.

SECONDARY OUTCOMES:
Awareness of health effects from smoking cigarettes | 4 weeks
  Awareness of health effects will be measured at 4 weeks by survey.
Awareness of cigarette smoke constituents | 4 weeks
  Awareness of constituents will be measured at 4 weeks by survey.
Quit attempts | Up to 4 weeks
  Quit attempt will be measured during the 4 weeks of the study, reported at either 2, 3, or 4 weeks. A quit attempt is defined as 24 hours without smoking.
Successful Quitting | 4 weeks
  Successful quitting will be defined as self-reported smoking on 0 of the past 7 days at 4 weeks.
Forgoing a cigarette | 4 weeks
  Forgoing a cigarette will be measured at 4 weeks as the frequency of butting out a cigarette or forgoing a cigarette in an effort to smoke less.
Perceived likelihood | 4 weeks
  Perceived likelihood of developing smoking-related health outcomes will be measured at 4 weeks by survey.
Frequency of conversations about health messages | 4 weeks
  Frequency of conversations with others about the health message on cigarette packs will be measured at 4 weeks by survey.
Negative affective reactions | 4 weeks
  Negative affect will be measured at 4 weeks by survey.
Cognitive elaboration | 4 weeks
  Cognitive elaboration (how much the participant reports thinking about the label) will be measured at 4 weeks by survey.

CONTACTS AND LOCATIONS:
Overall Officials: Noel Brewer, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Ewald & Wasserman Research Consultants, LLC, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brewer NT, Jeong M, Mendel JR, Hall MG, Zhang D, Parada H Jr, Boynton MH, Noar SM, Baig SA, Morgan JC, Ribisl KM. Cigarette pack messages about toxic chemicals: a randomised clinical trial. Tob Control. 2019 Jan;28(1):74-80. doi: 10.1136/tobaccocontrol-2017-054112. Epub 2018 Apr 13. PMID 29654122